CLINICAL TRIAL: NCT04886323
Title: Effect of Cold Atmospheric Plasma on Malassezia Folliculitis: a Randomized Controlled Trial
Brief Title: Effect of Cold Atmospheric Plasma on Malassezia Folliculitis
Acronym: ECAPMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Anhui Medical University (Other)
Collaborators: Hefei CAS Ion Medical and Technical Devices Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, Yang chunjun, Head of Dermatology, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YX2021-028
Record Dates: First submitted 2021-04-27; First posted 2021-05-14 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Malassezia Folliculitis
Keywords: Malassezia; Malassezia folliculitis; Cold atmospheric plasma; Pityrosporum folliculitis
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cold atmospheric plasma treatment group (Experimental): Patients are treated with a plasma device. Each treatment time was 3min per area based on the lesion size.The frequency of treatment is once a day. The duration of the treatment period is 2weeks.
  Interventions: Device: Cold atmospheric plasma treatment device
- Itraconazole capsules treatment group (Active Comparator): Patients are treated with Itraconazole capsules, 200mg a day.The duration of the treatment period is 2weeks.
  Interventions: Drug: Itraconazole Capsules

INTERVENTIONS:
Device: Cold atmospheric plasma treatment device — Treat with cold atmospheric plasma treatment device.
  Arms: cold atmospheric plasma treatment group
Drug: Itraconazole Capsules — Treat with Itraconazole capsules
  Arms: Itraconazole capsules treatment group

SUMMARY:
The cold atmospheric plasma may provide a new and effective method for the treatment of Malassezia folliculitis. The investigators conduct this randomized controlled trial to evaluate the effectiveness and safety of cold atmospheric plasma on Malassezia folliculitis. Participants entered this double-blind placebo-controlled trial will randomly assign to treatment with either cold atmospheric plasma or antifungal drugs. The differences of treatment effects of the two groups will be observed and compared.

DETAILED DESCRIPTION:
Malassezia folliculitis is a common disease of young and middle-aged people. It is an inflammatory disease caused by Malassezia infection. Generally, Topical or systemic use of antifungal drugs are the first choice for treatment but sometimes are limited due to adverse drug reactions and drug resistance. Cold atmospheric plasma has an inhibitory or killing effect on pathogenic microorganisms including fungi and has no obvious adverse damage to normal tissues. The investigators conduct this randomized controlled trial to study the effect of cold atmospheric plasma on Malassezia folliculitis, and evaluate its effectiveness and safety for Malassezia folliculitis. All data are recorded and compared after the end of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Patients are clinical presentation of Malassezia folliculitis in seborrheic areas.
* The diagnoses are mycologically verified by experienced laboratory technicians.
* Participants must be informed of the investigational nature of this study and be willing to provide written informed consent.

Exclusion Criteria:

* Combined with other serious systemic diseases.
* History of topical corticosteroids within 2 weeks or history of systemic corticosteroids within 1 month.
* History of immunosuppressive drugs within 1 month.
* History of topical antifungal medication within 2 weeks or systemic antifungal medication within 3 months.
* Pregnant and lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2023-12-17 (Actual)

PRIMARY OUTCOMES:
50% reduction in number of lesion | week 2
  proportion of subjects who achieve at least a 50% reduction in total number of lesions

SECONDARY OUTCOMES:
proportion of subjects in physician's global assessment. | week 2
  proportion of subjects who achieve a physician's global assessment 0 / 1.

CONTACTS AND LOCATIONS:
Overall Officials: Chunjun Yang, Study Chair — The Second Hospital of Anhui Medical University; Na Wang, Study Director — The Second Hospital of Anhui Medical University; Jingwen Wang, Principal Investigator — The Second Hospital of Anhui Medical University; Jing Gao, Principal Investigator — The Second Hospital of Anhui Medical University; Liyun Wang, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hald M, Arendrup MC, Svejgaard EL, Lindskov R, Foged EK, Saunte DM; Danish Society of Dermatology. Evidence-based Danish guidelines for the treatment of Malassezia-related skin diseases. Acta Derm Venereol. 2015 Jan;95(1):12-9. doi: 10.2340/00015555-1825. PMID 24556907
- [Background] VON Woedtke T, Schmidt A, Bekeschus S, Wende K, Weltmann KD. Plasma Medicine: A Field of Applied Redox Biology. In Vivo. 2019 Jul-Aug;33(4):1011-1026. doi: 10.21873/invivo.11570. PMID 31280189
- [Background] Wiegand C, Fink S, Hipler UC, Beier O, Horn K, Pfuch A, Schimanski A, Grunler B. Cold atmospheric pressure plasmas exhibit antimicrobial properties against critical bacteria and yeast species. J Wound Care. 2017 Aug 2;26(8):462-468. doi: 10.12968/jowc.2017.26.8.462. PMID 28795887
- [Background] Gao J, Wang L, Xia C, Yang X, Cao Z, Zheng L, Ko R, Shen C, Yang C, Cheng C. Cold atmospheric plasma promotes different types of superficial skin erosion wounds healing. Int Wound J. 2019 Oct;16(5):1103-1111. doi: 10.1111/iwj.13161. Epub 2019 Jun 17. PMID 31207094
- [Background] Parsad D, Saini R, Negi KS. Short term treatment of pityrosporum folliculitis with itraconazole. Indian J Dermatol Venereol Leprol. 1999 May-Jun;65(3):122-3. PMID 20921630
- [Background] Lee JW, Kim BJ, Kim MN. Photodynamic therapy: new treatment for recalcitrant Malassezia folliculitis. Lasers Surg Med. 2010 Feb;42(2):192-6. doi: 10.1002/lsm.20857. PMID 20166153
- [Background] Abdel-Razek M, Fadaly G, Abdel-Raheim M, al-Morsy F. Pityrosporum (Malassezia) folliculitis in Saudi Arabia--diagnosis and therapeutic trials. Clin Exp Dermatol. 1995 Sep;20(5):406-9. doi: 10.1111/j.1365-2230.1995.tb01358.x. PMID 8593718